CLINICAL TRIAL: NCT01830036
Title: RehaSleep Register - Prevalence of Sleep Apnea in Cardiac Rehabilitation
Acronym: RehaSleep
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-007
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Sleep Apnea
Keywords: cardiological treatment; sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quality of Life (SF12), 2-channel Polygraphy: cardiological treatment

SUMMARY:
Prevalence of sleep-related breath disturbance in patients in cardiac rehabilitation.

The aim of the register is to enable a better diagnosis and early treatment initiation in the context of secondary prevention. In addition to the prevalence, the further course of the patients shall be documented after hospital discharge to verify any gaps (sleep laboratory, therapy introduction) and emphasize the importance of rehabilitation and to examine the possibility of initiating therapy in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* terminal cardiac treatment in cardiac rehabilitation facility
* for example: Myocardial infarction, bypass surgery, stent implantation, valve replacement, ICD, CRT, pacemakers, heart failure

Exclusion Criteria:

* no informed consent form signed
* limited consent capacity (Dementia, addiction, psychosis)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment as part of the routine diagnostics using 2-channel polygraphic
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2011-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
cardiological treatment | April 2013
  all Patients who are admitted under a terminal cardiac treatment (myocardial infarction, bypass surgery, stent implantation, valve replacement, ICD, CRT) in a cardiac rehabilitation faciliy

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Krüger, Univ.-Prof., Principal Investigator — University Hospital Aachen, Medical Clinic I

REFERENCES:
- See also: juraforum online - sleep Apnea — http://www.juraforum.de/wissenschaft/schlafapnoe-herzpatienten-leiden-besonders-oft-unter-gefaehrlichem-schnarchen-434703